CLINICAL TRIAL: NCT03715036
Title: Point of Care Ultrasound Screening for Abnormal Fetal Growth During Routine Antenatal Visits: a Randomized Controlled Trial. MUNN (More Ultrasounds New gaiNs) Trial
Brief Title: Point of Care Ultrasound Screening for Abnormal Fetal Growth During Routine Antenatal Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #: 18-0023
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-06

CONDITIONS: Prenatal Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fundal height (No Intervention): Patients will have routine fundal height measurement
- Point-of-care US (Experimental): Patients will receive POC US for DVP and AC.
  Interventions: Diagnostic Test: Point-of-care US

INTERVENTIONS:
Diagnostic Test: Point-of-care US — The intervention includes reassuring the AC and DVP
  Arms: Point-of-care US

SUMMARY:
Abdominal circumference (AC) in the fetus is the single most useful indicator of fetal growth abnormalities. Measurement of AC as well as DVP do not require extensive training. Our objective is to evaluate if introduction of bedside ultrasound during routine antenatal visits to evaluate fetal AC and amniotic fluid DVP would decrease the false positive rates of fundal height measurement in diagnosing intrauterine growth abnormalities.

DETAILED DESCRIPTION:
The prior studies of routine ultrasound in low risk patients focused on the usual ultrasound evaluation which involves the use of advanced equipment and providers, including trained sonographers and physicians to perform and review the ultrasound, as well as a full examination with multiple fetal measurements and images. A number of recent analyses show that measurement of the abdominal circumference (AC) in the fetus is the single most useful indicator of fetal growth abnormalities. Measurement of AC as well as DVP do not require extensive training, long time to acquire, or expensive ultrasound machines. They can be easily performed in the office by providers who are specifically trained in obtaining these 2 measurements. Therefore, we intended to evaluate if introduction of bedside ultrasound during routine antenatal visits (point of care ultrasound or POC-US) to evaluate fetal AC and amniotic fluid DVP would decrease the false positive rates of fundal height measurement in diagnosing intrauterine growth abnormalities, and would improve the diagnosis of amniotic fluid volume and fetal growth deviations.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age ≥ 18 years and ability to give informed consent
2. Singleton gestation
3. Ultrasound examination that confirms or revises the EDD before 22 0/7 weeks of gestational age (ACOG Committee opinion 2017 dating)
4. Gestational age ≥ 24 weeks gestation

Exclusion Criteria:

1. Abnormal aneuploidy screening (1st trimester screening, 2nd trimester screening, integrated screening, NIPT)
2. Fetal chromosomal or genetic abnormalities
3. Fetal malformations or soft markers identified on fetal anatomy survey
4. Current pregnancy is a result of in vitro fertilization
5. Documented uterine bleeding after 24 weeks gestation. Unobserved self-reported bleeding with confirmed intact pregnancy on ultrasound after the bleeding episode is not an exclusion criteria.
6. Uterine/placental abnormalities including uterine malformations (i.e bicornuate uterus, didelpus uterus), abnormal placentation (placenta previa, accreta, percreta), uterine fibroids.
7. Cerclage in the current pregnancy
8. History of intrauterine fetal demise, small for gestational age, macrosomia or shoulder dystocia, or of traumatic delivery
9. Fetal isoimmunization or alloimmunization
10. History of medical complications such as:

    * Cancer (including melanoma but excluding other skin cancers)
    * Endocrine disease including thyroid disease (recently diagnosed or whose medication dose is not stable), adrenal disease, diabetes mellitus (pregestational and gestational).
    * Renal disease with altered renal function (creatinine > 0.9 or proteinuria)
    * Epilepsy or other seizure disorder
    * Any collagen disease (lupus erythematosus, scleroderma, etc.)
    * Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes)
    * Hematological disorder including alloimmune and isoimmune thrombocytopenia but excluding mild iron deficiency anemia (Hb > 9 gm/dl). Patients with sickle cell disease are excluded.
    * Chronic pulmonary disease including asthma requiring regular use of medication and active TB. An asthma inhaler used on an as needed basis (PRN) for a cold or an asthma attack is not considered regular use.
    * Heart disease except mitral value prolapse not requiring medication
    * Cardiovascular disorders: chronic hypertension
    * Liver disorders accounting for cholestasis
    * Infectious diseases: HIV, CMV, toxoplasmosis, parvovirus B19 Note that the aforementioned are just examples and any clinical indication for ultrasound examination after 24 weeks is an exclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Growth abnormalities rate | Up to 2 years
  To compare the false positive rates between clinical evaluation of uterine size by SFH versus POC-US evaluation of AC and DVP.

SECONDARY OUTCOMES:
MFM ultrasounds | Up to 2 years
  To compare fundal height (cm) versus bedside ultrasound on the overall rate of formal MFM ultrasound requests
Clinical evaluation | Up to 2 years
  To compare fundal height (cm) versus bedside ultrasound (abdominal circumference and Deep vertical pocket) on the prediction of birthweight < 10th percentile or > 90th percentile
Maternal and neonatal outcomes | Up to 2 years
  To compare maternal (emergency CD for non reassuring FHT, chorioamnionitis/post partum endometritis, wound infection/hematoma/seroma, PRBC transfusion, admission to the ICU, DVT/PE, maternal death) and perinatal (fetal death, neonatal death, Apgar score >< 4 at 5 min, neonatal seizures, umbilical-artery blood pH of 7.05 or less with a base deficit of 12 mmol per liter or more, intubation at delivery, neonatal encephalopathy) outcomes between strategy of clinical evaluation of uterine size versus bedside ultrasound (abdominal circumference and Deep vertical pocket)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Antonio, Principal Investigator — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Omere C, Goncharov DA, Pedroza C, La Rosa M, Munn M, Chiossi G, Longo M, Saad AF. Randomized trial of fundal height vs point-of-care ultrasound during routine antenatal visits. Am J Obstet Gynecol MFM. 2022 Mar;4(2):100563. doi: 10.1016/j.ajogmf.2022.100563. Epub 2022 Jan 13. No abstract available. PMID 35032696